CLINICAL TRIAL: NCT00599027
Title: An Exploratory Study of Mometasone Furoate Nasal Spray in Patients With Moderate-severe Persistent Allergic Rhinitis and Intermittent Asthma: Effects on the Quality of Life Evaluated With the Rhinasthma Questionnaire
Brief Title: An Exploratory Study of Nasonex in Patients With Moderate to Severe Persistent Allergic Rhinitis and Intermittent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05277
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone furoate nasal spray (Experimental): Mometasone furoate nasal spray (MFNS) 200 mcg once daily (two 50 mcg puffs per nostril) in the morning.
  Interventions: Drug: Mometasone furoate nasal spray (MFNS)
- Placebo nasal spray (Placebo Comparator): Placebo nasal spray once daily (two puffs per nostril) in the morning.
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Mometasone furoate nasal spray (MFNS) — Mometasone furoate nasal spray (MFNS) 200 mcg once daily (two 50 mcg puffs per nostril) in the morning.
  Other Names: Nasonex Nasal Spray
  Arms: Mometasone furoate nasal spray
Drug: Placebo nasal spray — Placebo nasal spray once daily (two puffs per nostril) in the morning.
  Other Names: Placebo
  Arms: Placebo nasal spray

SUMMARY:
The primary objective of this study is to explore the efficacy of Nasonex (mometasone furoate nasal spray) in comparison with placebo in improving the quality of life of subjects with moderate to severe persistent allergic rhinitis and intermittent asthma. A secondary objective is to evaluate the efficacy of Nasonex in relieving the subject's symptoms of allergic rhinitis and asthma.

DETAILED DESCRIPTION:
The primary objective is to explore the efficacy of mometasone furoate nasal spray (MFNS) in comparison with placebo in improving the quality of life of subjects with moderate to severe persistent allergic rhinitis and intermittent asthma as measured by the Rhinasthma Questionnaire (Global Summary Score). In addition, there are two secondary objectives. The first secondary objective is to evaluate the efficacy of MFNS in improving the quality of life of subjects with moderate to severe persistent allergic rhinitis and intermittent asthma as measured by the Rhinasthma Upper Airways Score, the Rhinasthma Lower Airways Score, and the Rhinasthma Respiratory Allergy Impact Score. The second secondary objective is to evaluate the efficacy of MFNS in relieving the subject's symptoms of allergic rhinitis and asthma as measured by the Total 5 Symptoms Score (T5SS) and the Global Symptom Score (T5SS+asthma symptoms) and by the use of rescue medication on demand.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients (≥18 and ≤ 75 years of age) of either sex
* Willingness to participate and comply with procedures by signing a written informed consent
* Moderate/severe persistent allergic rhinitis with a history of intermittent asthma from at least 2 years and actual asthma (symptoms in the last 4 weeks)
* To qualify at the randomization visit the daily average of the T5SS [(Morning-time T5SS + Evening-time T5SS)/2] had to be ≥ 6 in at least 4 days during the 1 week run-in period
* Positive (weal diameter >3 mm) skin prick test (SPT) and/or CAP-RAST (class II or higher) performed in the 6 months prior to the start of the trial were required for at least house dust mite and 1 pollen allergen (grass or Parietaria, IgE level >3.5 U/mL)
* All prior medication washout times had been observed
* Female volunteers of childbearing potential had to agree to use a medically accepted method of contraception or be surgically sterilized prior to screening, while receiving protocol-specified medication, and for 30 days after stopping the medication
* Negative urine pregnancy test
* Free of any clinically relevant disease that would have interfered with study evaluations
* Able to adhere to the dosing and visit schedules, and agree to record symptom severity scores and use of IMP and rescue medications in a daily diary

Exclusion Criteria:

* Female who was or intended to become pregnant during the study or within 12 weeks after study completion
* Nursing, or intended to be nursing during the study or within 12 months after study completion
* Taking medications prohibited during the study or had not complied with the requirements for the designated washout periods for any of the prohibited medications
* Anatomical abnormalities of the nose (turbinate hypertrophy, septal deviation, polyps)
* Acute or chronic sinusitis currently being treated with antibiotics and/or topical or oral decongestants
* Rhinitis medicamentosa
* Evidence of persistent asthma, or asthma with daytime and nighttime symptoms not controlled by short-acting beta2-adrenoceptor agonists
* Asthma requiring chronic use of inhaled or systemic corticosteroids
* Upper respiratory tract or sinus infection that required antibiotic therapy and had not had at least a 14-day wash-out period prior to the run-in period, or had a viral upper respiratory infection within 7 days prior to screening
* Dependence on nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids
* Undergoing a progressive course of immunotherapy (hyposensitization). Subjects on a regular maintenance schedule prior to the screening visit were eligible for study inclusion; however, subject could not receive hyposensitization treatment within 24 hours prior to any study visit
* Diagnosed of cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas)
* Concomitant medical problem
* Had any of the following clinical conditions: active or quiescent tuberculosis infection of the respiratory tract, untreated fungal, bacterial, systemic viral infections or ocular herpes simplex
* Smoked or had smoked within the previous 6 months
* Member of the staff, affiliated with, or family member of the staff personnel directly involved with this study
* Previously randomized into this study
* Any other clinically significant deviation from normal in the physical examination or medical history that could interfere with the study evaluation or affect subject safety
* In a situation or condition that could interfere with participation in the study
* Used any drug or device in an investigational protocol in the 30 days prior to visit 1
* Participating in other clinical studies
* Allergic or has sensitivity to the study drug or its excipients
* Compromised ability to provide informed consent
* History of non-compliance with medication or treatment protocols

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baiardini I, Villa E, Rogkakou A, Pellegrini S, Bacic M, Compalati E, Braido F, Le Grazie C, Canonica GW, Passalacqua G. Effects of mometasone furoate on the quality of life: a randomized placebo-controlled trial in persistent allergic rhinitis and intermittent asthma using the Rhinasthma questionnaire. Clin Exp Allergy. 2011 Mar;41(3):417-23. doi: 10.1111/j.1365-2222.2010.03660.x. Epub 2010 Dec 1. PMID 21121983

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Started | 26 | 25
Completed | 25 | 22
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Treatment Failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (13.42) | 43.0 (16.62) | 41.7 (14.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: The Change of the Rhinasthma Global Summary Score From Baseline to Endpoint After 28 Days of Treatment.
Description: To explore the efficacy of mometasone furoate nasal spray in comparison with placebo in improving the quality of life of subjects with moderate-severe PER and intermittent asthma as measured by the Rhinasthma Questionnaire (Global Summary Score). The Rhinasthma is a questionnaire that consists of 30 items and for each of them subjects had to indicate on a Likert scale (1=not at all; 5=very much) the degree of limitation or discomfort caused by each problem. Possible total best score = 150 and possible total worst score = 30.
Time Frame: Baseline and 28 days of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 26 | 25
units on a scale
  Baseline | 25.3 (10.03) | 26.7 (18.89)
  Endpoint after 28 days of treatment | -10.3 (7.15) | 0.4 (12.32)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Superiority or Other; p = 0.001, ANCOVA — Endpoint after 28 days of treatment; Overall treatment effect tested using F-test(alpha=0.05;two-sided). Diff between least square means of the 2 groups calculated with two-sided 95% C.I

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees not to publish or publicly present any interim results of the study without prior written consent of the sponsor. The PI further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication.